CLINICAL TRIAL: NCT01135316
Title: A Phase 4, Open-Label, Prospective Evaluation of the Incidence of Nephrogenic Systemic Fibrosis (NSF) in Patients With Moderate to Severe Kidney Disease Undergoing Magnetic Resonance Imaging (MRI) With Ablavar (Gadofosveset Trisodium) in Routine Clinical Practice
Brief Title: Prospective Evaluation of the Incidence of NSF in Patients With Kidney Disease Undergoing MR
Status: Completed | Type: Observational
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Other Study IDs: LMI-Ablavar-401
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Nephrogenic Systemic Fibrosis
Keywords: NSF, Ablavar, Kidney Disease, Magnetic Resonance Imaging (MRI),
MeSH Terms: conditions — Nephrogenic Fibrosing Dermopathy; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ablavar — One dose of Ablavar will be administered for use during a contrast MRI examination

SUMMARY:
Phase 4, open-label, two-year, prospective, multi-center, follow-up study conducted at up 15 sites in USA. Approximately 1,000 patients with moderate-to-severe CKD will be enrolled and followed for up to 24 months.

DETAILED DESCRIPTION:
Phase 4, open-label, two-year, prospective, multi-center, follow-up study will be conducted in up to 15 active sites in the United States. All patients will receive 1 dose of Ablavar as part of an MRI examination in their routine clinical management. Prior to undergoing an Ablavar MRI, patients will have a baseline serum creatinine test within 24 hours prior to Ablavar administration, will sign an Informed Consent (IC) form, will undergo a limited exam for skin abnormalities, and will undergo a brief medical history assessment on the day of and prior to Ablavar administration. A standardized NSF questionnaire will be administered to the patient at 48 (+ or -12) hours, 1 month (+ or - 1 week), 3 months (+ or - 2 weeks), 6 (+ or - 1) months, and 18 (+ or - 1) months post-dose. At 12 (+ or - 1) months, and at 24 (+ or - 1) months. Patients will return to the clinic for a limited examination for skin abnormalities and formal review of signs and symptoms suggestive of NSF.

ELIGIBILITY:
Inclusion Criteria:

Kidney Disease with GFR < 60 mL/min./1.73 m^2. Clinical Need to Receive an MRI with Contrast. Understand & Sign Informed Consent.

Exclusion Criteria:

History of known or suspected NSF. Has received any gadolinium based contrast agent within 12 months prior to enrollment.

Has a clinically significant skin disorder which may interfere with detection of cutaneous NSF manifestations.

Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data and achieving study objectives.

Is unable or unwilling to return for necessary office visits or follow up calls, and/or to be examined by a physician or undergo deep skin biopsy should the development of NSF be suspected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe kidney disease
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2009-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Nephrogenic Systemic Fibrosis | 24 months

SECONDARY OUTCOMES:
Incidence of Severe Adverse Events (SAEs) & Adverse Events (AEs) | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Simon P Robinson, PhD, Study Director — Lantheus Medical Imaging
Locations (2):
- United States (2):
  - Weill Cornell Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina